CLINICAL TRIAL: NCT03102931
Title: Switching to Low Oxidant Content Cigarettes in Adult Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, John P. Richie, Principal Investigator, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00006759; 5P50DA036107-02 (NIH)
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Nicotine; Oxidative Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Reduced ROS/RNS content products (Experimental): Participants will be given and asked to smoke research cigarettes for the first 4 weeks. For the final 4 weeks of the study they will be given and asked to smoke low ROS content cigarettes.
  Interventions: Other: Reduced ROS/RNS content products; Other: Typical to high (ROS/NOS) products

INTERVENTIONS:
Other: Reduced ROS/RNS content products — Participants will be given and asked to spoke only the cigarettes provided for them. Biosamples and surveys will be collected every 2 weeks throughout the study.
Other: Typical to high (ROS/NOS) products — Participants will be given and asked to spoke only the cigarettes provided for them. Biosamples and surveys will be collected every 2 weeks throughout the study.

SUMMARY:
The overall objective of this clinical study is to determine if smokers who switch from their usual high reactive oxygen and nitrous oxide species (ROS/NOS) products to a low ROS/NOS product exhibit increased or decreased levels of oxidative stress/damage, respectively.

DETAILED DESCRIPTION:
Researchers at Penn State Hershey are seeking healthy adult cigarette smokers between the ages of 21-65 who smoke at least 10 cigarettes a day for at least one year.

The aim of this study is to evaluate the effect of reduced oxidative/ nitrogen species (ROS/RNS) cigarettes compared to high ROS/RNS cigarettes.

Study participation lasts 8 weeks, with 5 study visits at the Hershey Medical Center. All eligible participants will be given Spectrum research cigarettes, provided free of charge, and will be asked to only smoke those cigarettes for the first four weeks of the study. Following that four-week period of time all participants will be given low ROS content cigarettes (American Spirit Dark Green or Pall Mall Red). Participants will be asked to smoke only these cigarettes for the final four weeks of the study, these cigarettes will also be provided to you free of charge.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65
* Smoke 10 cigarettes per day or more for at least one year
* Read and write in English
* Menthol and nonmenthol smokers
* Able to understand and provide consent to study procedures
* Plan to live in the local area for the next 3 months
* Women not pregnant or nursing and taking steps to avoid pregnancy
* No quit attempt in the last one months and not planning to quit in the next 3 months (ensuring stability of smoking)

Exclusion Criteria:

* Currently pregnant or nursing
* Unstable or significant medical conditions that affect oxidative stress, such as COPD, kidney failure, heart disease, stroke, cancer, tumors, lung or respiratory disease, diabetes, liver disease, autoimmune disorder, rheumatoid arthritis, infectious disease or fibromyalgia.
* Use of non-cigarette nicotine delivery
* History of difficulties providing blood samples: fainting, poor veins, anxiety, etc.
* Current or recent history of substance or alcohol abuse
* No more than seven alcoholic drinks a week, and/ or >two drinks a day
* Use of a high dose antioxidant supplement prior to 1 month
* Currently smoking cigarettes that will be used for the study (Pall Mall Red or American Spirit Dark Green)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
Biomarkers of oxidative stress | 8 weeks
  The primary endpoint is to assess whether levels of oxidative stress/damage increase or decrease when a smoker switches from a high ROS/NOS cigarette product to a low ROS/NOS product. The biomarkers that will be used to assess oxidative stress include: 8-0HdG, glutathionylated proteins, and urinary F,-isoprostanes cysteine and GSH.

SECONDARY OUTCOMES:
Antioxidant and nutrient levels in the blood | 8 weeks
  Secondary endpoints include measurements of nicotine exposure (urine or plasma cotinine).

CONTACTS AND LOCATIONS:
Overall Officials: John Richie, Ph.D, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this time we have no plan for sharing, however if need should arise, then sharing may be a possibility.